CLINICAL TRIAL: NCT01619501
Title: Dysregulation of the C/EBPa Pathway in Human Lung Cancer and Search for New Biomarkers and/or Therapeutic Targets
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/00117
Record Dates: First submitted 2012-04-04; First posted 2012-06-14 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The overall goal of this research is to enhance the investigators understanding of the pathways involved in lung cancer, and to identify new biomarkers and/or therapeutic targets. By comparing gene expression between normal lung tissue and tumors growing in lung-specific C/EBPa KO mice, the investigators have identified the Bmi-1 proto-oncogene as being abnormally upregulated in C/EBPa-deleted tumors. Subsequently, the investigators have validated this observation in human lung cancer, implicating the investigators KO mice are an effective discovery tool for lung cancer research. Through similar approaches, the investigators have already identified (Sonic Hedgehog, SHH), and plan to identify other pathways which are abnormally regulated in C/EBPa-/- tumors. In parallel, the investigators will proceed to define the clinical relevance of the SHH pathway and the other newly-discovered molecular aberrations, by analyzing their expression and correlate it to C/EBPa expression on the samples of patients with NSCLC at NUHS. If the investigators preliminary data on Bmi-1 will be confirmed, this proto-oncogene may generate useful correlates that could be used in diagnosis and treatment of lung cancer, as well as identify new prognostic/predictive markers in lung cancer. Similarly, SHH pathway-components may behave as potential biomarkers and therapeutic tools for C/EBPa-related lung cancers.

This proposal seeks to test the hypothesis that pathways which are dysregulated in lung tumors growing in a lung-specific C/EBPa KO model can be utilized as discovery tools to identify genes involved in human lung cancer pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

Patients with lung cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Archived samples from the Department of Pathology (for IHC, FISH) and the Tissue Repository (for fresh tumor samples) at NUHS
Sampling Method: Probability Sample
Dates: Start 2012-04; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Define the C/EBPa-Bmi-1 axis in human lung cancer
  Tissue microarrays will be created from the lung tumours. Only resection specimens will be used for TMA construction, and small, limited biopsies will not be used. Tissue punches of 1.5mm in diameter will be cut from the blocks (2 punches per tumour, 1 punch for normal lung). Hence the rest of the tumour block is not used, preserving most of the tumour tissue in the tissue blocks, for future diagnostic use.

SECONDARY OUTCOMES:
Validate the relevance of the C/EBPa-SHH pathway in human NSCLC
  We will stain the human lung cancer specimens with antibodies against Gli1 (the major effector of the SHH pathway), Patched-1, Patched-2 and Smoothened (the receptors of the pathway), Sonic, Indian and Desert Hedgehog (the ligands of the pathway), and Cyclin D, Cyclin E, and Myc (target genes of the pathway).Interestingly, the SHH pathway has been recently associated to primary cilia (PC), where its specific role is highly controversial. Genetic defects affecting PC result in a myriad of pathological instances, including lung pathologies
Identify new downstream targets of C/EBPa in murine lung cancer and test their involvement in human pathogenesis
  RNA microarray analysis will be performed by Dr. Levantini at the BIDMC (Tenen lab, Boston), to compare gene expression between C/EBPa-/- pulmonary tumors and the neighboring normal murine tissue. The mouse MOE430A gene chip from Affymetrix will be utilized, as recently published (Basseres et al., MCB 2006). Single cell suspension will be depleted by FACS for endothelial and hematopoietic markers (CD45, Ter119, CD31). Purified populations will then undergo cRNA synthesis followed by hybridization to the Affymetrix gene chips. The top 10,000 genes will be selected based on their ranking.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationa University Hospital, Singapore, Singapore